CLINICAL TRIAL: NCT02563119
Title: Characterization of Intestinal Microbiota in Healthy Subjects and Patients Before and After Bariatric Surgery Using Next Generation Sequencing Methods
Brief Title: Intestinal Microbiota in Patients Before and After Bariatric Surgery and Healthy Controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CBeglinger
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gastric Bypass Group (Active Comparator): Twenty morbidly obese patients undergoing gastric bypass surgery
  Interventions: Procedure: Gastric Bypass or Sleeve gastrectomy
- Sleeve Group (Active Comparator): Twenty morbidly obese patients undergoing sleeve gastrectomy
  Interventions: Procedure: Gastric Bypass or Sleeve gastrectomy
- Healthy controls (No Intervention): Thirty healthy, lean controls

INTERVENTIONS:
Procedure: Gastric Bypass or Sleeve gastrectomy
  Arms: Gastric Bypass Group; Sleeve Group

SUMMARY:
Studying obesity and metabolic syndrome attention is focused more and more on gut microbiota. In humans and animals, bariatric surgery (mainly gastric bypass surgery) lead to alterations of gut microbiota, which seem to be favourable. In this study the investigators aim to examine the effect of different bariatric procedures on composition of gut microbiota.

DETAILED DESCRIPTION:
The human gastrointestinal tract is home to an extremely numerous and diverse collection of microbes communities, collectively termed the "intestinal microbiota". This amazingly complex and poorly understood group of communities has an enormous impact on humans. Indeed, microbiota is considered to play a number of key roles in the maintenance of host health, including aiding digestion of otherwise indigestible dietary compounds, synthesis of vitamins and other beneficial metabolites, immune system regulation and enhanced resistance against colonization by pathogenic microorganisms. Conversely, the intestinal microbiota is also a potent source of antigens and potentially harmful compounds. Schematically, humans can be considered to exist in a state of natural balance with their microbial inhabitants. A shift in the balance of microbiota composition such that it may become deleterious to host health is termed "dysbiosis". Dysbiosis of the gut microbiota has been implicated in numerous disorders, ranging from intestinal such as inflammatory bowel diseases and colorectal cancer to disorders with more systemic effects such as diabetes, obesity, insulin resistance and steatohepatitis. The link between the microbes in the human gut and the development of obesity, cardiovascular disease and metabolic syndromes, such as type 2 diabetes, is becoming clearer but, because of the complexity of the microbial community, the functional connections are less well understood.

In humans and animals, bariatric surgery (mainly gastric bypass surgery) lead to alterations of gut microbiota, which seem to be favourable. In this study the investigators aim to examine the effect of different bariatric procedures on composition of gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* 30 healthy controls: BMI 18-30kg/m2 good general health
* 40 morbidly obese patients (BMI >35kg/m2) scheduled for either sleeve gastrectomy or gastric bypass surgery

Exclusion Criteria:

* Antibiotic therapy within the last 2 months before enrolment
* regular intake of proton pump Inhibitors (PPI)
* previous surgery on the gastrointestinal tract (appendectomy acceptable)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Characterization of of gut microbiome using next generation sequencing technology | six months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel,Division of Gastroenterology and Hepatology, Basel, Switzerland